# **INFORMED CONSENT FORM**

A Multicenter Phase II Study of Maintenance Belantamab Mafodotin (Blenrep®) After BCMA-Directed Chimeric Antigen Receptor T-cell Therapy in Patients With Relapsed and/or Refractory Multiple Myeloma

NCT05117008

IRB Approval Period: 12/14/2023 - 9/13/2024 Effective 12/14/2023

Clinical Interventions template - Version: December 1, 2020

IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

# Medical College of Wisconsin INTRODUCTION TO THE INFORMED CONSENT

IIT-CHHABRA-EMBRACE-MM: A Multicenter Phase II Study of Maintenance Belantamab Mafodotin (Blenrep®) after BCMA-Directed Chimeric Antigen Receptor T-Cell Therapy in Patients with Relapsed and/or Refractory Multiple Myeloma (RRMM)

Meera Mohan, MD
Department of Medicine
Medical College of Wisconsin
9200 West Wisconsin Avenue
Milwaukee WI 53226
414-805-6700

## **Definitions**

**CAR-T (Chimeric Antigen Receptor T-Cell) Therapy** – a special receptor created in the laboratory that is designed to bind to certain proteins on the cancer cell

**Biomarker –** something found in the blood, other fluids, or tissues that can be used to measure the progress of disease or how a treatment is working


Protocol Version: V3 v. 12/29/22

**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

#### **Purpose**

This project is being done to test the safety and effectiveness of a potential new treatment called Belantamab Mafodotin for subjects who have previously received at least three treatments, including CAR-T therapy.

#### Length

- 1. You will be in this research project for about up to 12 cycles or until your cancer gets worse.
- 2. We would also like to follow you in clinic visits and then for every 6 months to see how you are doing.

# **Procedures**

All subjects in this study will receive Belantamab Mafodotin. You will receive the study drug on Day 1 of every cycle. Each cycle is 56 days (8 weeks).

## List of visits:

Screening Visit(s)

- Total Number: about 1-3

- Total Time: about 4-10 hours each

Treatment Visits

- Total Number: about 12

- Total Time: about 3-6 hours each

Safety Follow-up Visit(s)

- Total Number: 1

- Total Time: about 4-6 hours

Pre-Progression Follow-up Visits

- Total Number: every 3 months until your cancer gets worse

- Total Time: about 2-4 hours each

Long Term Follow-up Visits (after progression)

- Total Number: every 6 months

- Total Time: about 1-4 hours each

## Risks

This is a brief list of the most commonly seen side effects. The *full consent form* after this introduction contains a more complete list of potential research risks.

#### **Belantamab Mafodotin risks:**

- Excess protein in the urine
- Eye problems: blurred vision, dry/itchy eyes, changes in vision, eye discomfort, difficulty seeing at night, inflammation or other changes of front part of eye
- Low number of blood cells called platelets
- Anemia
- Feeling sick to your stomach (nausea)
- Feeling tired (fatigue)
- Increase in liver function tests
- Fever
- Pneumonia, or other lung infection
- Cold or cold-like symptoms (upper respiratory tract infection)
- Low number of certain types of white blood cells called neutrophils (neutropenia) and lymphocytes (lymphopenia), which could increase the risk of infection. If you have a fever, please contact your study doctor immediately.
- Diarrhea
- Reactions from the infusion of Belantamab Mafodotin, usually happen within first 24 hours after the infusion. Symptoms may include flushing, chills, fever, difficulty breathing, rapid heartbeat, or a drop in blood pressure (feeling light-headed).


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

# Procedures that will occur at various visits:

# **Invasive Procedures**

Study drug administration (Belantamab Mafodotin), Blood collection, Bone marrow biopsy/aspirate, CT/PET/MRI scan

## **Non-invasive Procedures**

Physical examination and vital signs, Electrocardiogram (ECG), Echocardiogram (ECHO)/Multiple Gated Acquisition Scan (MUGA), Urine collection, Questionnaires, Skeletal survey

#### **Benefits**

We don't know if this project will help you. Your condition may get better but it could stay the same or even get worse.

## My Other Options

You do not have to join this project. Your other options may include:

- 1. Joining a different project
- 2. Routine care for this condition
- 3. Getting no treatment for this condition

If you have more questions about this project at any time, you can call Meera Mohan, MD at 414-805-6700.

If you have questions about your rights as a participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

## **CONSENT TO PARTICIPATE IN RESEARCH**

## A1. INTRODUCTION - WHY ARE WE ASKING YOU TO PARTICIPATE?

You are being invited to participate in this research because you have relapsed and/or refractory multiple myeloma and have previously received CAR-T therapy in addition to three other treatment regimens.

A total of about 45 people are expected to participate in this research nationally including about 10 at the Medical College of Wisconsin/Froedtert Hospital.

The Director of the project is Meera Mohan, MD in the Department of Medicine. A research team works with Meera Mohan, MD. You can ask who these people are.

GlaxoSmithKline (GSK), a drug company, is funding the research.

## **A2. DO I HAVE TO PARTICIPATE?**

You can decide whether to take part in this research or not. You are free to say yes or no. If you do not agree to join, or if you leave, you will not be penalized or lose any benefits that you had before starting the research project. Even if you join this project, you do not have to stay in it. You may stop at any time. Take as much time as you need to make your choice.

A research project is different from routine medical care in three ways: 1) there are extra risks that we will tell you about in this form; 2) you may have some extra medical tests and visits; 3) the research procedures, tests and visits follow a set plan that must be kept.

#### A3. WHY IS THIS PROJECT BEING DONE?

Current treatment regimens for multiple myeloma attempt to improve a patient's quality of life and prolong survival. These include stem cell transplant, chemotherapy, and other treatments which help to improve the immune system's function. However, over time many patients develop resistance to these treatments, and new treatment regimens are needed for these patients.

The purpose of this study is to test the safety and effectiveness of a potential new treatment called Belantamab Mafodotin for subjects who have previously received at least three treatments, including CAR-T therapy. Belantamab Mafodotin is investigational, meaning it is approved for other uses, but it is not approved by the FDA for use in this study.

Your condition may get better, but it could stay the same or even get worse. We hope the information from this study will help us develop a better treatment for multiple myeloma in the future.


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

#### **B1. WHAT WILL HAPPEN IF I PARTICIPATE?**

#### STUDY DRUGS

Belantamab Mafodotin is administered by intravenous (IV) infusion over a period of approximately 30 minutes. If you do not already have a port that has been surgically inserted, you will have a small catheter placed in a vein in your arm for the infusion. You will receive the infusion on Day 1 of every cycle lasting 56 days (8 weeks). The dosage will be determined based on your body weight and may change if you gain or lose weight.

You may receive pre-medication(s) up front, such as antihistamines, steroids, or pain relievers, to prevent drug reactions from happening, if you have side effects from similar drugs before or if your doctor think that it is needed in your case.

#### STUDY GROUPS

All subjects in this study will receive Belantamab Mafodotin.

#### STUDY VISTS

#### Screening

If you agree to participate in the study, you will sign this consent form before screening assessments are performed to see if you are eligible. Your study doctor or a member of the study team will let you know if you are eligible to participate in the study. If you are unable to participate in the study, the study doctor will discuss other treatment options with you.

#### **Treatment**

If you are eligible to participate, you will begin study drug treatment as described above. You will return to the clinic about once a week. Assessments to track your disease status and to monitor you for side effects will occur during the treatment visits. You will continue treatment with the study drug up to 12 cycles or until your cancer gets worse.

## Follow-up

After you stop study drug treatment, you will return to the clinic 70 days after your last dose for a Safety Follow-up visit to monitor for any side effects of the study drug.

If you stopped study drug treatment before your disease progressed, you will then be return to the clinic every 3 months for follow-up assessments to track the status of your disease. At progression, your medical record will be reviewed or you will be contacted every 6 months to see how you are doing.

If you stopped study drug treatment due to disease progression, your medical record will be reviewed or you will be contacted every 6 months to see how you are doing.


**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

MCW IRB

#### STUDY ASSESSMENTS

### Screening

You will need to have all or some of the following exams, tests, or procedures to find out if you can be in the study. Some of them are routine and may be done even if you do not join the study. If some of the tests were completed recently, they may not have to be repeated.

- Informed consent: Prior to any study-related procedures being performed, you will be required to voluntarily sign and date this consent form.
- Medical history: You will be asked about your health status, including previous treatments for your cancer
- Physical examination: You will receive a complete physical examination
- Eye Exam: You will have an eye exam performed to assess various parts of your vision
  - Visual Acuity: You will be asked to read different sized letters off a chart to test your vision (visual acuity). For this test, you will be asked to wear special glasses while different lenses are presented to you. We will test your visual acuity while you are wearing the lenses that allow you to read the most clearly
  - Eye Exam: A doctor may check your eyes using a low-powdered microscope with a bright light and magnifying lenses. As part of the eye exam, we may measure your intraocular pressure (the pressure inside your eye). To check your intraocular pressure, you will be given a numbing eye drop and then a special instrument will touch your eye for a few seconds to take a measurement. The doctor may also apply colored stains or dyes to the front of the eye to check for abnormalities of the surface layer of the eye (conjunctiva). The colored stain may be applied as a drop or using a sterile paper applicator dampened with eye wash or a numbing drop. If you have had a recent eye exam, we may be able to use information from your medical record instead of completing an eye exam during your study visit. We may also put drops in your eyes to dilate (or widen) your pupils.
  - o Additional examinations may be performed if the eye doctor thinks it is necessary
- Performance status: An assessment of your overall health and ability to perform daily tasks
- Medications: You will be asked about your current medications, including over-thecounter medications, vitamins, and herbal supplements
- Vital signs: Your blood pressure, heart rate, temperature, height, and weight will be checked
- Blood tests: Blood samples will be collected for
  - Blood cell counts, blood chemistry, clotting ability
  - Organ function
  - Active Hepatitis B and C infection

As part of the screening procedures, your blood will be tested for diseases that can be passed on to other people by transfusion, including Hepatitis B and C. If


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

certain tests are positive, we will inform you, and inform certain government health agencies as required by law. Results of your blood test will be released only to authorized persons as governed by Wisconsin law. A list of persons to be notified and reasons that will cause release of your blood test is available upon request. Results of the blood test will be released to the study team

- Pregnancy test (if you are a woman of childbearing potential)
- Indicators of your disease status
- Electrocardiogram (ECG) and Echocardiogram (ECHO)/Multiple Gated Acquisition Scan (MUGA): ECG and ECHO/MUGA will be performed to check the activity of your heart
- 24-hour urine and spot urine collections: Urine samples will be collected for indicators of your disease
- Whole-body PET/CT, CT, skeletal survey, and/or MRI: You will have a whole-body PET/ CT, CT, skeletal survey and/or MRI to assess your cancer
- Bone Marrow Biopsy and Aspirate: A bone marrow biopsy/aspiration is required and will be performed prior to the planned study treatment start date to assess disease status

#### **Treatment**

You will begin study drug treatment if the results of screening assessments show that you are eligible.

The following assessments will be performed at all treatment visits, unless noted.

- Medical history: You will be asked about your health status, including previous treatments for your cancer
- Physical examination: You will receive a complete physical examination
- Eye Exam: You will have an eye exam performed to assess various parts of your vision at all treatment visits except Cycle 1.
  - Visual Acuity: You will be asked to read different sized letters off a chart to test your vision (visual acuity). For this test, you will be asked to wear special glasses while different lenses are presented to you. We will test your visual acuity while you are wearing the lenses that allow you to read the most clearly
  - Eye Exam A doctor may check your eyes using a low-powdered microscope with a bright light and magnifying lenses. As part of the eye exam, we may measure your intraocular pressure (the pressure inside your eye). To check your intraocular pressure, you will be given a numbing eye drop and then a special instrument will touch your eye for a few seconds to take a measurement. The doctor may also apply colored stains or dyes to the front of the eye to check for abnormalities of the surface layer of the eye (conjunctiva). The colored stain may be applied as a drop or using a sterile paper applicator dampened with eye wash or a numbing drop. If you have had a recent eye exam, we may be able to use information from your medical record instead of completing an eye exam during your study visit. We may also put drops in your eyes to dilate (or widen) your pupils.


**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

- Additional examinations may be performed if the eye doctor thinks it is necessary
- Performance status: An assessment of your overall health and ability to perform daily tasks
- Medications: You will be asked about your current medications, including over-thecounter medications, vitamins, and herbal supplements
- Vital signs: Your blood pressure, heart rate, temperature, height, and weight will be checked
- Blood tests: Blood samples will be collected for
  - Blood cell counts, blood chemistry, clotting ability
  - Organ function
  - Pregnancy test (if you are a woman of childbearing potential)
  - Indicators of your disease status
- 24-hour urine and spot urine collections: Urine samples will be collected for indicators of your disease, at Cycle 2 and every other cycle thereafter
- Whole-body PET/CT, CT, skeletal survey, and/or MRI: You will have a whole-body PET/ CT, CT, skeletal survey and/or MRI to assess your cancer, at Cycle 7 only
- Bone Marrow Biopsy and Aspirate: A bone marrow biopsy/aspiration is required and will be performed prior to the planned study treatment start date to assess disease status, at Cycle 3 and Cycle 7
- Questionnaires: You will be asked to complete questionnaires about your ability to perform daily activities
- Bone marrow collection from diagnosis: We will analyze some of your stored bone marrow collected from your diagnosis, at Cycle 1 only

#### Follow-up

# Safety Follow-up Visit

The following assessments will be performed 70 days after you stop study drug treatment:

- Medical history: You will be asked about your health status, including previous treatments for your cancer
- Physical examination: You will receive a complete physical examination
- Eye Exam: You will have an eye exam performed to assess various parts of your vision.
  - Visual Acuity: You will be asked to read different sized letters off a chart to test your vision (visual acuity). For this test, you will be asked to wear special glasses while different lenses are presented to you. We will test your visual acuity while you are wearing the lenses that allow you to read the most clearly
  - Eye Exam: A doctor may check your eyes using a low-powdered microscope with a bright light and magnifying lenses. As part of the eye exam, we may measure your intraocular pressure (the pressure inside your eye). To check your


**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

intraocular pressure, you will be given a numbing eye drop and then a special instrument will touch your eye for a few seconds to take a measurement. The doctor may also apply colored stains or dyes to the front of the eye to check for abnormalities of the surface layer of the eye (conjunctiva). The colored stain may be applied as a drop or using a sterile paper applicator dampened with eye wash or a numbing drop. If you have had a recent eye exam, we may be able to use information from your medical record instead of completing an eye exam during your study visit. We may also put drops in your eyes to dilate (or widen) your pupils.

- Additional examinations may be performed if the eye doctor thinks it is necessary
- Performance status: An assessment of your overall health and ability to perform daily tasks
- Medications: You will be asked about your current medications, including over-thecounter medications, vitamins, and herbal supplements
- Vital signs: Your blood pressure, heart rate, temperature, height, and weight will be checked
- Blood tests: Blood samples will be collected for
  - Blood cell counts, blood chemistry, clotting ability
  - Organ function
  - Pregnancy test (if you are a woman of childbearing potential)
  - Indicators of your disease status
- 24-hour urine and spot urine collections: Urine samples will be collected for indicators of your disease
- Whole-body PET/CT, CT, skeletal survey, and/or MRI: You will have a whole-body PET/ CT, CT, skeletal survey and/or MRI to assess your cancer
- Bone Marrow Biopsy and Aspirate: A bone marrow biopsy/aspiration is required and will be performed to assess disease status
- Questionnaires: You will be asked to complete questionnaires about your ability to perform daily activities

# Pre-Progression Follow-up Visits

You will return to the clinic every 3 months from your Safety Follow-up visit until your cancer gets worse to monitor your health. The following assessments will be performed at each Pre-Progression Follow-up visit:

- Medical history: You will be asked about your health status, including previous treatments for your cancer
- Physical examination: You will receive a complete physical examination
- Performance status: An assessment of your overall health and ability to perform daily tasks


# **Informed Consent for Research**


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

- Medications: You will be asked about your current medications, including over-thecounter medications, vitamins, and herbal supplements
- · Height and weight: Your height and weight will be checked
- Blood tests: Blood samples will be collected for
  - Blood cell counts, blood chemistry, clotting ability
  - Organ function
  - Pregnancy test (if you are a woman of childbearing potential)
  - Indicators of your disease status
- 24-hour urine and spot urine collections: Urine samples will be collected for indicators of your disease

If the study doctor thinks it is necessary, you will continue to have eye exam visits every 3 months until 1 year from the end of the study treatment. Additional examinations may be performed if the eye doctor thinks it is necessary.

#### Long-Term Follow-up

After your cancer gets worse, we will contact you every 6 months to see how you are doing.

## STUDY SAMPLES FOR RESEARCH

We would also like to collect samples during the study to be used for future research. These samples are required to participate in the main study. The samples will be used to analyze different biomarkers. A biomarker is something found in the blood, other fluids, or tissues that can be used to measure the progress of disease or how a treatment is working.

The following samples will be collected at the visits listed below:

Bone marrow aspirate (about 5-10 mL at each time point)

- Screening
- Cycle 3 Day 1
- Cycle 7 Day 1
- 70 days post-last dose safety visit or progression, whichever is earlier
- Bone marrow that was collected from your diagnosis

Blood (about 15 mL of blood at each time point)

- Screening
- Cycle 3 Day 1
- Cycle 7 Day 1
- 70 days post-last dose safety visit or progression, whichever is earlier


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

#### **GENETIC TESTING**

In this project, we will do genetic testing on your biospecimens. This will be collected at the time points listed in the "STUDY SAMPLES FOR RESEARCH" heading above. Genetic testing will be done because researchers would like to better understand the mechanisms of how the study drug affects your multiple myeloma.

This genetic testing is for research only. The purpose is not to discover information that could be used to change your medical care, make or change your diagnosis, or advise you on your risk of diseases.

The biospecimens collected for this part of the project will be coded, which means they will be labeled with numbers and/or letters instead of information that could identify you. Only the research team will be able to link the code to you. The samples will also be labeled with date of collection, which could potentially be used to identify you. The research team will make every effort to protect the information and keep it confidential, but it is possible that an unauthorized person might see it. Depending on the kind of information being collected, it might be used in a way that could embarrass you.

It is against federal law (Genetic Information Nondiscrimination Act, or GINA) for health insurance companies to deny health insurance, or large employers to deny jobs, based on your genetic information. But the same law does not protect your ability to get disability, life, or long-term care insurance. If you have questions, you can talk to the research doctor about whether this could apply to you.

You will not be given your genetic test results.

## **B2. HOW LONG WILL I BE IN THE PROJECT?**

You will continue treatment with the study drug up to 12 cycles or until your cancer gets worse.

After you stop study drug treatment, you will return to the clinic 70 days after your last dose for a Safety Follow-up visit to monitor for any side effects of the study drug.

If you stopped study drug treatment before your disease progressed, you will then be return to the clinic every 3 months for follow-up assessments to track the status of your disease. At progression, your medical record will be reviewed or you will be contacted every 6 months to see how you are doing.

If you stopped study drug treatment due to disease progression, your medical record will be reviewed or you will be contacted every 6 months to see how you are doing.

## **B3. CAN I STOP BEING IN THE PROJECT?**

You are free to withdraw from the project at any time. If you leave, your regular medical care will not change. If you are thinking about leaving, please tell the research doctor.

The research doctor can tell you about the effects of stopping, and you and the research doctor can talk about what follow-up care would help you the most.


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

12/14/2023

**EFFECTIVE** 

MCW IRB

You might be asked to come back for one more visit to check your health.

The research doctor may take you out of this project at any time. This would happen if:

- They think it is in your best interest.
- You do not follow the project rules.
- The whole project is stopped.

If this happens, the research doctor will tell you.

## **B4. ARE THERE ANY SPECIAL INSTRUCTIONS WHILE I AM IN THE PROJECT?**

You must attend all of the study appointments. If you have to miss an appointment, you must reschedule with the study doctor or staff.

You must tell the study doctor about any medicines you are currently taking or may take during the course of the study (e.g., prescription, vitamins, over the counter, herbal supplements etc.), as some of these may need to be stopped/reduced.

You must not wear contact lenses while participating this study. If you are experiencing discomfort in your eyes, please talk to your doctor about the use of preservative-free artificial tears or cooling eye masks.

Please discuss with your doctor if you plan to receive any vaccines, including the COVID-19 vaccine.

You should not breastfeed a baby while you are participating in the study and for 3 months after the last dose of study drug.

#### C1. WHAT HEALTH RISKS OR PROBLEMS CAN I EXPECT FROM THE PROJECT?

There are risks to taking part in any research project. There is a risk that you may get a drug that does not help your condition or may make it worse. There also may be problems (side effects) we do not know about yet, from the drug itself, or how it combines with other drugs you are taking. If we learn about new important side effects, we will tell you.

We watch everyone in the project for problems (side effects). You need to tell the research doctor or a member of the research team immediately if you experience any problems, side effects, or changes in your health. In an emergency, call 911.

# **C2. RISKS OF STUDY DRUG**

The research drug itself may cause problems (side effects). Side effects may be mild or very serious. Some can last a long time or never go away.

Many go away soon after you stop taking the drugs. Drugs can affect individuals in different ways. Complications of some of the side effects below may lead to life-threatening events, possibly resulting in death.


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

The side effects that other people have experienced so far with the study drug are:

#### **Belantamab Mafodotin**

Belantamab Mafodotin is an approved drug in the European Union, United Kingdom, Switzerland, Singapore, Hong Kong, and Israel with ongoing clinical development; therefore, not all of its side effects are known at this time. As of 27 February 2023, over 1,600 people with MM have received Belantamab Mafodotin across all ongoing and completed clinical studies.

Some common side effects reported with Belantamab Mafodotin are described below.

## Eye Problems

Some participants who have received Belantamab Mafodotin in clinical studies developed problems in the front part of the eve called the cornea. Sometimes the changes can only be observed by an eye doctor during eye examination, and they do not result in any symptoms. Those changes might be more frequent in patients who had problems with dry eye prior to treatment with Belantamab Mafodotin. Some patients, however, develop symptoms related to Belantamab Mafodotin. The symptoms could range from a feeling of dryness in the eye to more severe symptoms, like blurry vision or changes in your eyesight, that could affect your ability to see things clearly and may affect your reading ability or difficulty in driving. A few people have developed eye sores. These effects typically go away if the study drug is held and the dose reduced upon re-start, but please discuss with your study doctor if you have questions. In severe cases, sores can develop on the eye, possibly with infection. If untreated this could potentially lead to scarring which may permanently affect your eyesight. If you experience new eye symptoms (such as pain or irritation, blurry vision, or feeling like something is in your eye), you should urgently seek medical attention by an eye care specialist. Your eyes will be examined repeatedly during the study, as it is important to monitor the effects of Belantamab Mafodotin on your eyes. If you develop problems with your eyesight or other problems with your eyes, do not drive or operate heavy machinery until you have had your eyes examined by an eye care specialist.

## Abnormal Bruising and Bleeding

Belantamab Mafodotin can decrease the number of blood cells called platelets, which help to clot your blood. Symptoms of low platelets counts (called thrombocytopenia) can include abnormal bruising of your skin, bleeding for longer than usual after your blood has been drawn, or bleeding from your nose or gums. In some cases, the bleeding can occur from other areas of your body. Bleeding may be serious, or life threatening and may require a transfusion. Your study doctor will closely monitor your platelets by checking your blood tests before you start your treatment and regularly during the study.

## Infusion-related reactions

Some people may have allergic-like reactions when they receive an infusion of Belantamab Mafodotin. These usually develop within minutes or hours but can develop up to 24 hours after your dose is given. It is a reaction to the drug being a foreign protein, and you may have flushing, chills, fever, problems with breathing, feeling like your heart is racing or a drop in blood pressure (which may cause you to feel dizzy, light-headed or like you're going to faint). You will usually spend an hour after your dose to check whether you will develop these symptoms but if you experience any of these symptoms at any time contact your study doctor immediately.


**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

# Inflammation of the lungs

Some people who have received Belantamab Mafodotin experienced inflammation of the lungs which can cause cough, shortness of breath and difficulty breathing, and in some cases, death. It is not certain if Belantamab Mafodotin causes the inflammation or not. If you experience new or worsening breathing problems like cough or shortness of breath with an unknown cause, contact your study doctor immediately.

#### Excess protein in the urine

Some people receiving Belantamab Mafodotin have developed excess levels of protein (called albumin) in the urine, which can sometimes be a sign of a kidney disorder. Your study doctor will closely monitor protein levels in your urine regularly during the study. If your urine looks foamy or frothy or if you notice new swelling or more swelling than usual in your feet, legs or other parts of your body, contact your study doctor immediately.

# Side Effects

The side effects described below are from 95 patients with RRMM who received at least one dose of Belantamab Mafodotin at doses of 2.5 mg/kg.

The most common side effects occurring in more than 20% of people (20 or more out of 100 people) were:

- Eye problems: blurred vision, dry/itchy eyes, changes in vision, eye discomfort, difficulty seeing at night, inflammation or other changes of front part of eye.
- Low number of blood cells called platelets (thrombocytopenia), which may cause bleeding and easy bruising. Bleeding may be serious, or life threatening and may require a transfusion.
- Having fewer red blood cells than normal (anemia)
- Feeling sick to your stomach (nausea)
- Feeling tired (fatigue)
- Increase in liver function tests
- Fever (if you have a fever, please contact your study doctor immediately)
- Pneumonia, or other lung infection
- Cold or cold-like symptoms (upper respiratory tract infection)
- Low number of certain types of white blood cells called neutrophils (neutropenia) and lymphocytes (lymphopenia), which could increase the risk of infection. If you have a fever, please contact your study doctor immediately.
- Diarrhea
- Reactions from the infusion of Belantamab Mafodotin, usually happen within first 24 hours after the infusion. Symptoms may include flushing, chills, fever, difficulty breathing, rapid heartbeat, or a drop in blood pressure (feeling light-headed).


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

Other common side effects seen in 1% to 10% of subjects (between 1 to 10 out of 100 people) were:

- Other eye problems: eye irritation, abnormal sensitivity of the eyes to light, and cores on the eyes possibly with infection.
- Increased albumin, a type of protein in the urine, (albuminuria)
- An increase in an enzyme released into the blood when muscle is damaged (creatine phosphokinase)
- Vomiting

In another study which is testing Belantamab Mafodotin in combination with two medicines already approved for the treatment of RRMM, called Lenalidomide and Dexamethasone, two patients who had low neutrophil counts developed serious infections which led to death.

**Embryo-fetal toxicity:** Belantamab Mafodotin may harm an unborn baby. You must have negative pregnancy tests to continue in the study if you are a woman who can have children.

Fertility: Belantamab Mafodotin treatment may affect men and women's ability to have children.

There may be other side effects that may happen that are not known now. For example, all drugs can cause an allergic reaction in some participants. Certain problems can become worse if not treated quickly. Call the study doctor right away if:

- You feel very tired or faint
- You feel pain or sick in your stomach and you do not want to eat
- You bruise easily or develop itching
- You have yellow eyes or skin, or dark urine
- You become confused.

#### C3. OTHER RISKS OF THIS RESEARCH PROJECT

Other procedures that are part of the research also involve some risks:

### Intravenous (IV) Drug Administration

It is recommended that the study drug is given into a vein in the arm. There is a risk that the study drug could leak outside the vein. If that happens, the drug could leak into the surrounding tissue and cause considerable irritation, and even tissue damage. The nurses and doctors will take every precaution to prevent leaks from the peripheral line, but there is still a risk that the tissue around the injection site could become damaged if it comes into contact with the study drug. Immediately tell the study doctor or nurse if you feel a burning sensation or irritation at the injection site any time during or after being given the study drug.

#### **Blood Draws:**

Blood draws are necessary to monitor the disease being treated as well as the side effects of the treatment. However, by participating in the study you may require a higher frequency of blood draws that would be performed if your doctor was treating you with standard,


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

nonexperimental therapies. Risks associated with blood draws include pain, itching, and, more rarely, anemia, fainting and dizziness.

# Electrocardiogram (ECG)

An ECG is a simple and painless test that detects and records the electrical activity of your heart. Soft adhesive patches the size of a quarter (called electrodes) will be attached to the skin of the chest, arms, and legs. You will be requested to lie still for a few minutes while a machine records the electrical signals. Rarely, localized rash or skin irritation may occur where the electrode patches are placed. These reactions are typically temporary.

# **Echocardiogram (ECHO)**

During the echocardiogram, electrodes will be placed onto your chest to allow for an ECG to be performed. Then a transducer (a device that looks like a computer mouse) will be applied. You may feel slight pressure on your chest from the transducer. In addition, you may be asked to breathe in a certain way or to rest on your side during the test.

## Multiple Gated Acquisition Scan (MUGA)

A MUGA scan takes images of the beating heart to see how well your heart is pumping blood. A small amount of radioactive material will be injected into your vein and bind to your red blood cells (blood cells that carry oxygen throughout your body) in order for the special camera to take pictures of how the blood moves through your heart. You will be asked to lie very still during this scan, because any movement can cause the images to be blurry. There may be some discomfort from having to lie still during the length of the procedure. Allergic reactions to the radioactive material are rare but may occur. The injection of the radioactive material may cause some slight discomfort.

#### Bone marrow biopsy or aspirate

Your study doctor will explain the risks associated with collecting the bone marrow biopsy and/or aspiration. Having a biopsy or aspiration performed may cause some pain, bruising, redness, inflammation, bleeding, low blood pressure, swelling and/or infection at the site of the biopsy or aspiration.

#### **PET Scan**

Positron emission tomography (PET) is a type of imaging test that uses a small amount of radioactive material injected into your vein to see how cells or tissues are functioning. It is combined with a CT scan (3D x-ray) in one machine so doctors can better see the structures the PET agent goes to.

Before the scan, you will have to follow preparation instructions including not eating for 6 hours before the test. After the PET agent is injected, you will wait 45-60 minutes before being scanned. The scan will take several minutes, and you must lie still during that time.

## CT Scan

CT scans use x-rays to create an image. If frequent CT scans are performed, the cumulative amount of radiation involved could be concerning. People who have a small but increased radiation exposure may have the risk of cancer development in later life. However, there is considerable uncertainty regarding the risk estimates for low levels of radiation exposure from the CT scans you will undergo.


**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

# Skeletal survey X-ray

An X-ray exposes your body to radiation. The amount of radiation you get from an X-ray is small, and from skeletal survey X-rays it is usually equal to 4–6 months of background radiation.

#### MRI Scan

MRI, which uses a large magnet instead of x-rays to take pictures of your body, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish.

The MRI may require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm people who have metal in their bodies (pacemakers, neurostimulators, certain clips, or staples from surgery). It may cause problems with devices, such as pacemakers. If you have metal in your body or a pacemaker, you should not have an MRI. Your study doctor will discuss with you whether you should have a MRI scan with a contrast agent based on your health status.

## **Eye Exam Procedures**

## Eye Exam

The lights used by the doctor for the eye exam are bright and may be uncomfortable, but they are not expected to harm your eyes. Intraocular pressure testing can rarely cause minor scratching to the front of the eye. Since you will be given numbing drops before this test, it is important to avoid rubbing your eyes for at least fifteen minutes after receiving the drops, since small particles or dust could scratch the front of your eye without you noticing any pain. Colored stains used for the exam may cause mild irritation and may cause your eye to look discolored temporarily. If you wear contact lenses and put them in while the stain is still present, the stain may discolor your contact lens

#### **Pupil Dilation**

Dilating drops may sting temporarily when they are placed in your eyes. While your eyes are dilated, you will likely experience blurred vision, difficulty focusing, and sensitivity to light. You may also experience a headache or watering of the eyes. The effect of the dilating drops lasts several hours. Very rarely (less than 1% of the time), you may have redness, discomfort, or an allergic reaction to the drops that are used to dilate the pupil. This is generally not serious and can be treated if it occurs. Some types of glaucoma (i.e., angle-closure glaucoma) may be made worse by dilating drops in some people, but this can also be treated.

## **Quality of Life Questionnaires**

The answers that you give are confidential, but there is always a risk that your answers will be read by people who should not read your personal information. You may also feel uncomfortable completing some of the assessments.


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

## **Privacy and Confidentiality**

Another risk may be loss of confidentiality. Every effort will be made to keep your research records confidential but we cannot guarantee it. Depending on the kind of information being collected, if your research information were accidentally seen, it might be used in a way that could embarrass you or affect your ability to get insurance. If you have questions, you can talk to the project director about whether this could apply to you.

#### **C4. REPRODUCTIVE RISKS**

## Risks to subjects who could become pregnant

We do not know if the drug causes harm to a baby, so we do not want anyone who might be pregnant to enter the project.

You should not become pregnant or nurse a baby while in this project. You must tell the research doctor right away if you think you are pregnant. You will be asked to have a pregnancy test to be sure you are not pregnant at the start of the project, during the project, and at the end of the project.

You may not donate eggs during your participation in the project or for 4 months after stopping the drug.

If you become pregnant during the project, the research drug will be stopped for safety reasons. If you become pregnant while you are taking this experimental drug or within 4 months after you have stopped taking it, we ask that you inform the research doctor immediately. The research doctor will ask you for written permission to obtain information from you or your obstetrician on your pregnancy and the health of the baby.

## Risks to a subject who could father a child and the subject's partner(s)

If you and your partner(s) are able to become pregnant, one or both of you must use some form of effective birth control, because it is unknown if the drug could affect a baby. You must tell the research doctor right away if you think your partner is pregnant.

You may not donate sperm during your participation in the project or for 6 months after stopping drug.

If you think you have gotten your partner pregnant while you are taking this experimental drug or within 6 months after you have stopped taking it, we ask that you inform the research doctor immediately. At that time, the research doctor will ask permission of your partner for the use and disclosure of health information regarding the pregnancy. Your partner will be asked to sign a separate consent form and can choose to do this or not. Your partner will be asked to sign this form to allow your research doctor to contact your partner's obstetrician to collect information on the progress of the pregnancy and its outcome. The research doctor will make this information available to the sponsor for safety monitoring.

#### Birth control methods for all subjects

Check with the research doctor about the birth control methods needed for this project and how long to use them. Some methods might not be good enough for this project. If you are having sex that could lead to pregnancy, you should use one form of highly effective birth control while you are in this project.


**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

12/14/2023

**EFFECTIVE** 

**MCW IRB** 

## This may include:

- Not having vaginal sex (abstinence)
- Taking birth control pills orally
- Having birth control shots or patches such as Depo-Provera
- Surgical sterilization (hysterectomy/tubal ligation or vasectomy)
- Limiting sexual activity to a partner who has undergone surgical sterilization
- Use of an intrauterine device (IUD)
- Use of diaphragm with contraceptive jelly
- Use of condoms with contraceptive foam
- Use of diaphragm with condoms ("double barrier")

Subjects able to become pregnant should use birth control for 4 months after stopping the study drug.

Subjects able make their partners pregnant should use birth control for 6 months after stopping the study drug.

#### C5. ARE THERE ANY BENEFITS TO TAKING PART IN THE PROJECT?

We don't know if this study will help you. Your condition may get better, but it could stay the same or even get worse. We hope the information from this study will help us develop better treatments multiple myeloma.

#### D1. ARE THERE ANY COSTS TO BEING IN THE PROJECT?

Most of the medical care that you will receive in this project is considered routine care for your condition and would be recommended whether or not you join the project. Costs for routine care will be billed to you or your insurance carrier. For routine clinical care, you will be responsible for paying any copayment, coinsurance, or deductible that is required by your insurance carrier.

Activities / costs that are part of the project will not be billed to you or your insurance company. These are: the study drug, Belantamab Mafodotin; all Eye exams required for this study; the ECG at screening; the ECHO/MUGA done at screening; labs not part of your normal care that are drawn or collected for research purposes; and the processing and shipping of research samples.

Some insurers will not pay for drugs, tests or hospitalization that are part of research, so check with your insurer before you join this project. If you have questions regarding costs, please contact Dr. Mohan.

If you participate in this research, the costs of any necessary emergency medical treatment in the event of a research-related injury will be billed to you or your health insurance.

## D2. WILL I BE PAID FOR PARTICIPATING IN THE PROJECT?

There is no payment for being in this project.


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

Sponsor, other researchers, or research companies may patent or sell products, discoveries and data or information that result from this research. Neither Sponsor nor Dr. Mohan will pay you if this happens. You will not receive any payment or commercial rights for products, data, discoveries, or materials gained or produced from your biospecimens.

## D3. WHAT OTHER HEALTHCARE CHOICES DO I HAVE?

You do not have to join this project. You are free to say yes or no. If you do not join this project, your research doctor can discuss other healthcare choices with you.

Your other choices may include:

- Routine care for your type of cancer, including other FDA-approved therapies for relapsed/refractory multiple myeloma. Belantamab Mafodotin is also available to you as standard of care approved by the FDA if you have progressive myeloma.
- Joining a different research project

The research doctor can explain both the possible benefits and the risks of other options that are available to you.

## D4. WILL I BE GIVEN NEW INFORMATION ABOUT THE PROJECT?

If we learn any important new information about the drugs that might change your mind about being in the project, we will tell you about it right away. You can then decide if you want to stay in the project.

When research biospecimens are collected and analyzed, there is the chance of finding something clinically relevant. There may be benefits to learning such results (such as early detection and treatment of a medical condition), but there are risks as well (such as feeling worried about a finding for which no treatment is required or appropriate).

The results from the biospecimens we collect in this research study are not the same quality as what you would receive as part of your health care, so you will not be informed of any clinically relevant research findings. The results of your research biospecimens will not be placed in your medical record.

#### D5. WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THE PROJECT?

Emergency medical treatment for injuries directly related to your participation in this research project will be provided to you. You or your health insurance will be billed for the costs of this emergency treatment. MCW will decide on a case by case basis if they will reimburse you or your insurer for emergency treatment costs. If your research-related injury requires medical care beyond this emergency treatment, you or your insurer will be responsible for the costs of this follow-up care.

At this time, there is no plan for any additional financial payments.

If you believe that you have been injured because of your participation in this project, contact the research doctors right away. Contact information: Meera Mohan, MD, 414-805-6700


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

Nothing in this consent form affects any legal rights you may have nor does it release the investigator, the sponsor, the institution, or its agents from liability for negligence.

#### D6. WHO CAN ANSWER MY QUESTIONS ABOUT THE PROJECT?

- If you have more questions about this project at any time, you can call Meera Mohan, MD at 414-805-6700.
- If you have questions about your rights as a research participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.

## E. PERMISSION TO COLLECT, USE AND SHARE HEALTH INFORMATION

# E1. What health information will be collected and used for this project?

To be in this research project, the research team needs your permission to access, collect and use some of your health information. If you say no, you cannot be in the project. This information may come from questions we ask, forms we ask you to fill out, or your medical record, as described below. We will only collect and use information needed for the project.

The protected health information (PHI) originates from services you will or have received at one or more of the following locations: the Medical College of Wisconsin (MCW); Versiti, Inc.; Children's Hospital of Wisconsin (CHW); any Froedtert Health Affiliate- Froedtert Hospital (FH), Inc.; Froedtert Menomonee Falls Hospital; Froedtert West Bend Hospital; Froedtert & The Medical College of Wisconsin Community Physicians Clinics, Inc. (FMCWCP); the West Bend Surgery Center, LLC; and the Froedtert Surgery Center, LLC.

## The health information to be collected and used for this project is:

- Past and present medical records to document relevant pre-existing conditions
- Records about your Study visits and results of tests done during the study
- Records about phone calls made as part of this research
- Research records

# E2. Who will see the health information collected for this project?

The only MCW/Froedtert Hospital employees allowed to handle your health information are those on the research team, those on the Institutional Review Board (IRB) and those who check on the research activities to make sure the hospital's rules are followed.

If the costs of any necessary emergency medical treatment in the event of a research-related injury are billed to your health insurance, your health information may need to be disclosed to the insurer for billing purposes.

The research team may share your information with people who don't work at MCW/Froedtert Hospital because they planned, pay for, or work with us on this project. The federal Privacy Rule may no longer protect your health information once it leaves MCW/Froedtert Hospital. For this project, we plan to share information with those doctors, researchers or government representatives working with us on this project at the institutions or companies listed here:


**Informed Consent for Research** 


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

Florence Healthcare, Inc.

- The study sponsor and its research partners
- Doctors and healthcare professionals at other sites taking part in the study
- Companies that fund the study
- Government agencies in the U.S., such as the Food and Drug Administration (FDA), National Cancer Institute (NCI), and National Institutes of Health (NIH)

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

- Other federal and state agencies, such as the Office of Human Research Protections, (OHRP)
- Those required by law who monitor research data

Because this project involves the use of drugs and/or devices, the FDA also has the right to inspect all project records.

We may record your research information, including results of tests and procedures done for research, in your Froedtert Hospital and/or Medical College of Wisconsin medical record. As a result, this research information may be seen by people allowed to see your medical records for healthcare operations or treatment, by those you allow to see your medical records by giving written permission, and by others when required by law.

We will not use your personal health information for a different project without your permission or the permission of a hospital research review board (IRB). Once all personal identification is removed from your health information and/or biospecimens, the information and/or biospecimens may be used for future research or distributed to another investigator for future research without additional informed consent from you or your legally authorized representative. The information might also be used or released for other purposes without asking you. Results of the project may be presented in public talks or written articles, but no information will be presented that identifies you.

## E3. What are the risks of sharing this health information?

One risk of taking part in a research project is that more people will handle your personal health information collected for this project. The research team will make every effort to protect the information and keep it confidential, but it is possible that an unauthorized person might see it. If you have questions, you can talk to the research doctor about whether this could apply to you.

## E4. How long will you keep the health information for this project?

If you sign this form, we plan to keep your information without any end-date in case we need to check it again for this project.

#### E5. Can I cancel my permission to share this health information?

If you change your mind later and do not want us to collect or share your health information, you need to send a letter to Meera Mohan, MD at

Department of Medicine Medical College of Wisconsin 9200 West Wisconsin Avenue Milwaukee WI 53226


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

The letter must say that you have changed your mind and do not want the researcher to collect and share your health information. At that time, we will decide that you cannot continue to be part of the project. We may still use the information we have already collected.

## E6. Access to records

You may not be able to see, or copy, your project-related health information until after the project has been completed; otherwise, it could affect the study.

#### F1. FOR MORE INFORMATION ABOUT THE PROJECT

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can look up this project by referring to the ClinicalTrials.gov number (NCT05117008) or by asking the research team for a printed copy.


IRB Protocol Number: PRO 42276

IRB Approval Period: 12/14/2023 - 9/13/2024

**EFFECTIVE** 

12/14/2023

**MCW IRB** 

## **CONSENT TO PARTICIPATE**

# By signing my name below, I confirm the following:

- I have read (or had read to me) this entire consent document.
   All of my questions have been answered to my satisfaction.
- The project's purpose, procedures, risks and possible benefits have been explained to me.
- I agree to let the research team use and share the health information and other information gathered for this project.
- I voluntarily agree to participate in this research project. I agree to follow the procedures as directed. I have been told that I can stop at any time.

**IMPORTANT:** You will receive a signed and dated copy of this consent form. Please keep it where you can find it easily. It will help you remember what we discussed today.

| Subject's Name please print | Subject's Signature | Date |
|---|---|---|
| Name of Witness, if applicable please print | Signature of Witness | Date |
| Rationale for Use of Witness | | • |
| ☐ Subject has limited/no literacy | ☐ Sponsor requirement | |
| ☐ Subject has limited English | ☐ Other | |
| proficiency | | |
| ☐ Subject has limited/no vision | | |
| * Name of person discussing/<br>obtaining consent please print | Signature of person discussing/obtaining consent | Date |


<sup>\*</sup> A member of the research team trained and authorized by the Principal Investigator to act on her/his behalf in obtaining informed consent according to the protocol. The Principal Investigator is responsible and accountable for the research project.